CLINICAL TRIAL: NCT03496987
Title: Vacuum vs Manual Drainage During Unilateral Thoracentesis: A Randomized Trial
Brief Title: Vacuum vs Manual Drainage During Unilateral Thoracentesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1511016858; P30AG021342 (NIH)
Record Dates: First submitted 2018-04-04; First posted 2018-04-12 (Actual); Results first posted 2018-08-31 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Pleural Effusion; Pleural Diseases; Thoracic Diseases
Keywords: Pleural Effusion; Pleural Drainage; Thoracentesis
MeSH Terms: conditions — Pleural Effusion; Pleural Diseases; Thoracic Diseases

STUDY DESIGN:
Intervention Model Description: Patients are randomly assigned immediately before performing the procedure to either of the two investigational arms: manual drainage or vacuum bottle drainage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Drainage (No Intervention): Patients undergo drainage of pleural fluid via manual (syringe) system
- Vacuum Bottle Drainage (Experimental): Patients undergo drainage of pleural fluid via a vacuum bottle system (evacuated cylinder)
  Interventions: Device: Vacuum Bottle Drainage

INTERVENTIONS:
Device: Vacuum Bottle Drainage — Patients undergo drainage via vacuum bottles
  Other Names: Evacuated Cylinder
  Arms: Vacuum Bottle Drainage

SUMMARY:
The purpose of this study is to determine if there are any differences in terms of safety, pain, or drainage speed between thoracenteses via manual drainage vs vacuum suction.

DETAILED DESCRIPTION:
Patients with pleural effusions routinely undergo thoracentesis in which a catheter is placed into the pleural space to remove the fluid both for diagnostic and therapeutic reasons. In this setting, large amounts (often liters) of fluid are removed to palliate the patient's symptoms of breathlessness.

Thoracentesis is the most commonly performed and least invasive method to remove pleural fluid. These frequently performed using a catheter drainage system where a small, flexible temporary catheter is inserted over a needle into the pleural cavity. After insertion of catheter into the pleural space, the operator has two drainage system options: 1. Manual drainage via syringe-pump that connects to drainage bag or 2. Drainage into a vacuum bottle. Both are routinely performed in almost every hospital in the United States.

Pleural pressure (Ppl) is determined by the elastic recoil properties of the lung and chest wall. Normal pleural pressure is estimated to be -3 to -5 cm H20 at functional residual capacity. During drainage of pleural fluid, negative pressure is applied either via syringe during manual drainage or via vacuum using vacuum drainage bottle. Hypothetically more negative pressure can translate to increased perception of pain or visceral pleural injury.

Two techniques (manual vs vacuum drainage) are used based on the operator preference and both are standard of care. To our knowledge there is no head to head comparison of these two available systems of drainages during thoracentesis of pleural effusions. Knowing if one is superior to the other will aid future clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral therapeutic thoracentesis

Exclusion Criteria:

* Patients with a history of prior significant pleural or lung based procedures/surgeries (not a simple thoracentesis)
* Prior enrollment in this study
* Patients ability to comprehend and consent to this procedure and clearly communicate any pain or other symptoms that arise from this procedure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan T Puchalski, MD, MEd, Principal Investigator — Yale University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puchalski JT, Argento AC, Murphy TE, Araujo KL, Pisani MA. The safety of thoracentesis in patients with uncorrected bleeding risk. Ann Am Thorac Soc. 2013 Aug;10(4):336-41. doi: 10.1513/AnnalsATS.201210-088OC. PMID 23952852
- [Background] Jones PW, Moyers JP, Rogers JT, Rodriguez RM, Lee YC, Light RW. Ultrasound-guided thoracentesis: is it a safer method? Chest. 2003 Feb;123(2):418-23. doi: 10.1378/chest.123.2.418. PMID 12576360
- [Background] Havelock T, Teoh R, Laws D, Gleeson F; BTS Pleural Disease Guideline Group. Pleural procedures and thoracic ultrasound: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii61-76. doi: 10.1136/thx.2010.137026. No abstract available. PMID 20696688
- [Background] Seneff MG, Corwin RW, Gold LH, Irwin RS. Complications associated with thoracocentesis. Chest. 1986 Jul;90(1):97-100. doi: 10.1378/chest.90.1.97. PMID 3522123
- [Background] Roth BJ, Cragun WH, Grathwohl KW. Complications associated with thoracentesis. Arch Intern Med. 1991 Oct;151(10):2095-6. doi: 10.1001/archinte.151.10.2095a. No abstract available. PMID 1929699
- [Background] Raptopoulos V, Davis LM, Lee G, Umali C, Lew R, Irwin RS. Factors affecting the development of pneumothorax associated with thoracentesis. AJR Am J Roentgenol. 1991 May;156(5):917-20. doi: 10.2214/ajr.156.5.2017951.
- [Background] Heidecker J, Huggins JT, Sahn SA, Doelken P. Pathophysiology of pneumothorax following ultrasound-guided thoracentesis. Chest. 2006 Oct;130(4):1173-84. doi: 10.1378/chest.130.4.1173. PMID 17035453
- [Background] Josephson T, Nordenskjold CA, Larsson J, Rosenberg LU, Kaijser M. Amount drained at ultrasound-guided thoracentesis and risk of pneumothorax. Acta Radiol. 2009 Jan;50(1):42-7. doi: 10.1080/02841850802590460. PMID 19052935
- [Background] Feller-Kopman D, Walkey A, Berkowitz D, Ernst A. The relationship of pleural pressure to symptom development during therapeutic thoracentesis. Chest. 2006 Jun;129(6):1556-60. doi: 10.1378/chest.129.6.1556. PMID 16778274
- [Background] BEECH RD. Practical system for thoracentesis using the blood donor set. J Am Med Assoc. 1951 Aug 25;146(17):1597. doi: 10.1001/jama.1951.63670170006011d. No abstract available. PMID 14861005
- [Background] ALBERTSON HA, LEAVITT D, GAMBLE JR. A simple method for doing a thoracentesis using a plasma-collecting vacuum bottle. J Thorac Surg. 1954 Nov;28(5):544-5. No abstract available. PMID 13212859
- [Background] Puchalski JT, Argento AC, Murphy TE, Araujo KL, Oliva IB, Rubinowitz AN, Pisani MA. Etiologies of bilateral pleural effusions. Respir Med. 2013 Feb;107(2):284-91. doi: 10.1016/j.rmed.2012.10.004. Epub 2012 Dec 7. PMID 23219348
- [Background] Petersen WG, Zimmerman R. Limited utility of chest radiograph after thoracentesis. Chest. 2000 Apr;117(4):1038-42. doi: 10.1378/chest.117.4.1038. PMID 10767236
- [Background] Kelil T, Shyn PB, Wu LE, Levesque VM, Kacher D, Khorasani R, Silverman SG. Wall suction-assisted image-guided therapeutic paracentesis: a safe and less expensive alternative to evacuated bottles. Abdom Radiol (NY). 2016 Jul;41(7):1333-7. doi: 10.1007/s00261-016-0634-x. PMID 27315094
- [Background] Alraiyes AH, Kheir F, Harris K, Gildea TR. How Much Negative Pressure Are We Generating During Thoracentesis? Ochsner J. 2017 Summer;17(2):138-140. No abstract available. PMID 28638284

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inpatients, who were awake, consentable, and undergoing unilateral thoracentesis
Period: Overall Study
Arm/Group | Manual Drainage | Vacuum Bottle Drainage
Started | 49 | 51
Completed | 49 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Drainage | Vacuum Bottle Drainage | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (16.2) | 65.6 (15.5) | 67 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 23 | 29 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 49 | 51 | 100

OUTCOME MEASURES:

1. Primary Outcome: Pain Change
Description: Difference in pain between pre-procedural pain and during drainage pain as measured as the difference between a pre-procedural NPSS pain score (range from 0 (no pain) to 10 (maximum pain)). This was asked again during drainage and the difference between the two was recorded. The values ranged from -10 to 10 (with a more negative number representing a decrease in pain and a more positive number representing an increase in pain)
  The scale used is called The Numeric Pain Rating Scale. With ratings from 0-10. Zero is the least amount of pain experienced while 10 is the worst pain possible.
Time Frame: 5-20 minutes
Population: 1 patient was excluded from analysis from the Vacuum Bottle Drainage arm from the original 51 enrolled because of a technical problem with the drainage system (not a complication).
Measure: Mean (Standard Deviation); unit: Pre-post NPRS Pain Scale Score
Arm/Group | Manual Drainage | Vacuum Bottle Drainage
Number analyzed (Participants) | 49 | 50
Pre-post NPRS Pain Scale Score | 0.53 (1.7) | 1.43 (2.7)

2. Secondary Outcome: Time of Drainage
Description: Actual time of drainage in seconds for each patient.
Time Frame: 5-20 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Manual Drainage | Vacuum Bottle Drainage
Number analyzed (Participants) | 49 | 50
seconds | 498.5 (386.5) | 318.6 (193)

3. Secondary Outcome: Number of Patients Who Had an Early Termination of Procedure
Description: Patients who had procedure termination prior to complete evacuation of the pleural contents (usually as a result of refractory pain or another symptom that the patient perceived).
Time Frame: 5-20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Manual Drainage | Vacuum Bottle Drainage
Number analyzed (Participants) | 49 | 51
Participants | 1 | 8

4. Secondary Outcome: Number of Patients Who Had a Complication as a Result of the Procedure
Description: Any complications that occur as a direct result of the procedure. We tracked patients for 7 days after the procedure to capture any complications (which is typical clinical practice)
Time Frame: <7 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Manual Drainage | Vacuum Bottle Drainage
Number analyzed (Participants) | 49 | 50
Participants
  Pneumothorax | 0 | 3
  Hemothorax | 0 | 1
  Clinically Significant Pulmonary Edema | 0 | 1

5. Secondary Outcome: Etiology of Effusion
Description: Clinical etiology of effusion
Time Frame: <7 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Manual Drainage | Vacuum Bottle Drainage
Number analyzed (Participants) | 49 | 50
Participants
  Malignant | 13 | 8
  Paramalignant | 7 | 2
  Heart Failure | 7 | 8
  Hepatic Hydrothorax | 3 | 5
  Post-Cardiothoracic Procedure | 13 | 17
  Parapneumonic | 3 | 2
  Unknown | 3 | 8

6. Secondary Outcome: Volume of Effusion
Description: Volume of effusion drained (in mL)
Time Frame: <20 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliters
Arm/Group | Manual Drainage | Vacuum Bottle Drainage
Number analyzed (Participants) | 49 | 50
milliters | 1023 (674) | 1143 (775)

7. Secondary Outcome: Laterality of Effusion
Description: Laterality of effusion (left or right)
Time Frame: <20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Manual Drainage | Vacuum Bottle Drainage
Number analyzed (Participants) | 49 | 51
Participants
  Left | 17 | 23
  Right | 32 | 28

ADVERSE EVENTS:
Time Frame: 1 month following procedure
Arm/Group | Manual Drainage | Vacuum Bottle Drainage
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/49 | 5/51
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Manual Drainage (N=49) | Vacuum Bottle Drainage (N=51)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) — Pneumothorax as a result of the procedure
Clinically Significant Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Clinically Significant Pulmonary Edema requiring ventilatory support
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Hemothorax (or bleeding in the thoracic cavity as a result of the procedure)

LIMITATIONS AND CAVEATS:
This was a single center study with a modest patient size. There was heterogeneity between the two arms of the study which limits interpretation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2015-11-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT03496987/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT03496987/SAP_001.pdf
  • Informed Consent Form (2015-11-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT03496987/ICF_002.pdf